CLINICAL TRIAL: NCT05917197
Title: Assessing the Impact of Social Media on the Development of Anorexia Nervosa in Undergraduate Students-A Cross Sectional Study From a Developing Country
Brief Title: Impact of Social Media on the Development of Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: Jinnah Sindh Medical University (Other)
Responsible Party: Principal Investigator, Areeba Ismail, Areeba Ismail, Jinnah Sindh Medical University
Other Study IDs: 2021-576
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: The Focus of Study Were the Medical Students Whose Eating Behaviors Were Studied

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical students
  Interventions: Other: survey based information

INTERVENTIONS:
Other: survey based information — Only survey based information collected

SUMMARY:
The study involves the recruitment of medical students from all government medical colleges of Karachi,Pakistan. The sample size was 214. The study is a cross sectional study that requires the participants to fill out an online questionnaire after giving an informed consent online.

DETAILED DESCRIPTION:
The study involves the recruitment of medical students from all government medical colleges of Karachi, Pakistan. The sample size was 214. The study is a cross sectional study that requires the participants to fill out an online questionnaire after giving an informed consent online.The questionnaire contained 15 items related to their social media use and its impact on their body image and eating behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Medical students of Karachi
* All should be aged 18 to 25 years
* Both genders included

Exclusion Criteria:

* Non consenting participants
* Those who donot have access to social media

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical students of Karachi
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Social media use | 6 months
  Instagram usage was more as compared to other social media sites

CONTACTS AND LOCATIONS:
Overall Officials: Areeba Ismail, Principal Investigator — Jinnah Sindh Medical University
Locations (1):
- Sindh, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared amongst other researchers